CLINICAL TRIAL: NCT07157254
Title: A Phase 2, Open-label, Basket Study Investigating the Safety and Efficacy of GTX-102 in Adult and Pediatric Subjects With Deletion- or Nondeletion-type Angelman Syndrome
Brief Title: A Safety and Efficacy Study of GTX-102 in Subjects With Deletion- or Nondeletion-type Angelman Syndrome (AS)
Acronym: Aurora
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTX-102-CL210; 2024-519393-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Subprotocol A GTX-102 (Experimental): Participants with deletion-type Angelman syndrome, ≥1 to <4 years of age will receive increasing doses of GTX-102 via intrathecal (IT) injection until the target dose is achieved. Dosing occurs every 3 months (Q3M) thereafter.
  Interventions: Drug: GTX-102
- Subprotocol B GTX-102 (Experimental): Participants with paternal uniparental disomy (UPD)/imprinting center defect (ICD) Angelman syndrome, ≥4 to <18 years of age will receive increasing doses of GTX-102 via IT injection until the target dose is achieved. Dosing occurs Q3M thereafter.
  Interventions: Drug: GTX-102
- Subprotocol C GTX-102 (Experimental): Participants with all genotypes of Angelman syndrome, ≥18 to <65 years of age will receive increasing doses of GTX-102 via IT injection until the target dose is achieved. Dosing occurs Q3M thereafter.
  Interventions: Drug: GTX-102
- Subprotocol D GTX-102 (Experimental): Participants with mutation-type Angelman syndrome, ≥4 to <18 years of age will receive increasing doses of GTX-102 via IT injection until the target dose is achieved. Dosing occurs Q3M thereafter.
  Interventions: Drug: GTX-102
- Subprotocol D No Intervention then GTX-102 (Experimental): Participants with mutation-type Angelman syndrome, ≥4 to <18 years of age will receive no treatment during the initial period. At the end of the no treatment period, participants will receive increasing doses of GTX-102 via IT injection until the target dose is achieved. Dosing occurs Q3M thereafter.
  Interventions: Other: No intervention; Drug: GTX-102

INTERVENTIONS:
Other: No intervention — During the no treatment period participants do not receive any study drug
  Arms: Subprotocol D No Intervention then GTX-102
Drug: GTX-102 — antisense oligonucleotide
  Other Names: apazunersen

SUMMARY:
The main goal of the study is to evaluate the safety and efficacy of GTX-102 in participants with Angelman syndrome.

DETAILED DESCRIPTION:
This basket study is designed to evaluate safety and efficacy of GTX-102 in participants with Angelman syndrome across genotypes and age groups. The study consists of subprotocols A, B, C and D. All subprotocols are open-label and follow the same design which includes a Screening, Loading and Maintenance period. Subprotocols A, B and C are single arm only. In subprotocol D, participants are randomized 2:1 to a GTX-102 group or a No Treatment group. The No Treatment group follows the same schedule of events as all other groups after completion of the No Treatment period. Participants from all the subprotocols have the option to continue treatment in a long-term extension study following their end of study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parent(s) or legal guardian(s)
2. Males and females of the following ages and genotypes at time of informed consent:

   1. Subprotocol A: ≥ 1 to < 4 years of age with a genetically confirmed diagnosis of deletion-type Angelman syndrome
   2. Subprotocol B: ≥ 4 to < 18 years of age with a genetically confirmed diagnosis of UPD/ICD Angelman syndrome
   3. Subprotocol C: ≥ 18 to < 65 years of age with a genetically confirmed diagnosis of Angelman syndrome, any genotype
   4. Subprotocol D: ≥ 4 to < 18 years of age with a genetically confirmed diagnosis of mutation-type Angelman syndrome
3. Weight ≥ 8 kg at Screening Visit
4. Platelet count, prothrombin time / international normalized ratio, and partial thromboplastin time < 1.5x the upper limit of normal and platelets > 75,000 cells/mm3 at the Screening Visit
5. Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, and all study procedures, including lumbar puncture (LP) procedure, magnetic resonance imaging (MRI) and tolerating anesthesia without intubation
6. From the time of informed consent through to at least 6 months after the final dose of GTX-102, females of childbearing potential who are sexually active must use highly effective contraception or abstinence. Males are able to participate if they agree to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the study and for at least 3 months after the final dose of GTX-102

Exclusion Criteria:

1. Any change in medications or diet/supplements intended to treat symptoms of Angelman Syndrome (eg, sleeping aids, antiseizure medications, supplements, dietary change including ketogenic or low-glycemic index diet, other) within the month prior to the Screening Visit (excluding weight-based adjustments)
2. Any condition that creates an increased risk of unsuccessful lumbar puncture
3. Current or expected concomitant use of drugs that increase the risk of bleeding (eg, heparin, low molecular weight heparin, platelet inhibitors)
4. Known hypersensitivity to GTX-102 or its excipients or required premedication that, in the judgment of the Investigator, places the subject at increased risk for adverse effects
5. Presence or history of any condition, lab abnormality, or infection that, in the judgment of the Investigator, would interfere with study participation, pose undue safety risk, or would confound interpretation of results
6. Pregnant or breastfeeding or planning to become pregnant (self or partner) at any time during the study
7. Use of any investigational product or investigational medical device within 6 months or 5 half-lives prior to the Screening Visit, or any prior use of gene therapy or an ASO regardless of length of time since last use
8. Concurrent participation in any interventional study

Ages: 1 Year to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Subprotocol A/B/C/D: Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs), Severe Events, and Events Related to Investigational Product, Procedure, and Premedication | Up to Day 506
Subprotocol A Only: Bayley-4 Cognitive Without Caregiver Input Raw Score Change from Baseline at Day 338 | Baseline, Day 338
Subprotocol B/D Only: Multidomain Responder Index (MDRI) Net Response at Day 338 | Baseline, Day 338
  The following assessments will be included to calculate the MDRI net response: Bayley-4 Cognitive and Receptive Communication, Aberrant Behavior Checklist- Community (ABC-C) Hyperactivity/Noncompliance (H/N), Angelman Severity Assessment (ASA) Sleep, ASA Gross Motor. For each assessment a meaningful score difference (MSD) is defined. A single net response score per participant will be derived accordingly, and a summary measure of net response will then be calculated across all participants.
Subprotocol C Only: MDRI Net Response at Day 338 | Baseline, Day 338
  The following assessments will be included to calculate the MDRI net response: Vineland-3 Expressive and Receptive Communication, ABC-C Irritability, ASA Gross Motor. For each assessment a meaningful score difference (MSD) is defined. A single net response score per participant will be derived accordingly, and a summary measure of net response will then be calculated across all participants.

SECONDARY OUTCOMES:
Subprotocol A/B/D Only: Change From Baseline at Day 338 in Bayley-4 Receptive Communication Raw Score | Baseline, Day 338
Subprotocol A/B/D Only: Change From Baseline at Day 338 in Bayley-4 Gross Motor Raw Score | Baseline, Day 338
Subprotocol B/D Only: Change From Baseline at Day 338 in Bayley-4 Cognitive Raw Score | Baseline, Day 338
Subprotocol B/C/D Only: Change From Baseline at Day 338 in Vineland-3 Receptive Communication Raw Score | Baseline, Day 338
Subprotocol B/C/D Only: Change From Baseline at Day 338 in Vineland-3 Expressive Communication Raw Score | Baseline, Day 338
Subprotocol B/D: Change From Baseline at Day 338 in Aberrant Behavior Checklist-Community (ABC-C) Hyperactivity/Noncompliance Raw Score | Baseline, Day 338
Subprotocol B/D Only: Change From Baseline at Day 338 in Angelman Severity Assessment (ASA) Sleep Rating | Baseline, Day 338
Subprotocol B/C/D Only: Change From Baseline at Day 338 in ASA Gross Motor Rating | Baseline, Day 338
Subprotocol C Only: Change From Baseline at Day 338 in ABC-C Irritability Raw Score | Baseline, Day 338

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (22):
- United States (9):
  - Clinical Trial Site, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Kansas City, Missouri
  - Rare Disease Research, Hillsborough, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - UT Health Austin, Austin, Texas
  - Carum Research Inc., Dallas, Texas
- Clinical Trial Site, Pilar, Buenos Aires, Argentina
- Brazil (2):
  - Clinical Trial Site, Curitiba, Paraná
  - Clinical Trial Site, Santa Cecília, Porto Alegre
- France (2):
  - Clinical Trial Site, Marseille
  - Clinical Trial Site, Paris
- Clinical Trial Site, Ramat Gan, Israel
- Italy (3):
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Rome
- Portugal (2):
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- United Kingdom (2):
  - Clinical Trial Site, London
  - Clinical Trial Site, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy Website — https://www.ultrarareadvocacy.com/conditions-we-study/angelman-syndrome-as/
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/